CLINICAL TRIAL: NCT06280079
Title: Efficacy, Safety, and Tolerability of Ultra-high-caloric, Fatty Diet (UFD) in Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Ultra-high-caloric, Fatty Diet in ALS
Acronym: LIPCAL-ALS II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Albert Christian Ludolph, Prof., Prof. Dr., University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIPCAL-ALS II 1.1
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; High-caloric, high-fat nutrition; Survival; Randomized controlled trial
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultra-high-caloric fatty diet (Experimental): ultra-high-caloric, high-fat, fluid nutritional supplement oral intake of 4 times 35 ml per day in addition to normal food intake, corresponding to +630 kcal and +70g fat per day
  Interventions: Dietary Supplement: Ultra-high-caloric fatty diet
- Placebo (Placebo Comparator): placebo, fluid nutritional supplement oral intake of 4 times 35 ml per day in addition to normal food intake, corresponding to +50 kcal and +3,5g fat per day
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ultra-high-caloric fatty diet — 100% fat (70g), saturated fatty acids 7,5g, monounsaturated fatty acids 42,6g, polyunsaturated fatty acids 19,9g, long-chain fatty acids 100%, ratio omega-6 to omega-3 fatty acids 5:1, protein 0g, carbohydrates 0g, fiber 0g
  Arms: Ultra-high-caloric fatty diet
Other: Placebo — <5% fat (<3,5g), protein 0g, carbohydrates 0g, fiber 0g
  Arms: Placebo

SUMMARY:
This study aims at evaluating efficacy and tolerability of an ultra-high-caloric, fatty diet (UFD) compared to placebo in patients with amyotrophic lateral sclerosis (ALS).

DETAILED DESCRIPTION:
ALS is a fatal neurodegenerative disease, leading to progressive paralysis of voluntarily innervated muscles and to death caused by respiratory failure after a mean disease duration of 2-4 years.The proposed study aims at improving survival of ALS patients by targeting metabolic parameters. ALS patients feature an intrinsic hypermetabolism as signified by an increased resting energy expenditure, which significantly contributes to progressive weight loss and cachexia. The extent of weight loss is an independent prognostic factor for survival in ALS. It has been shown that survival of ALS mice can be prolonged by applying a high-caloric nutrition. Furthermore, ALS patients feature distinct alterations of lipid metabolism, and various studies suggest a protective effect of high triglyceride serum levels.

In the precursor-study LIPCAL-ALS-I, a randomized, placebo-controlled, multicenter trial, evaluating the effects of a high-caloric fatty diet (HCFD), the primary endpoint (survival in the whole study population) was missed. However, post-hoc analysis revealed showed that HCFD (1) increased survival and reduced weight loss in normal to fast-progressing patients (patients with a functional decline measured by ALS Functional Rating Scale Revised) above the median at baseline; p=0.02), (2) slowed down functional decline (measured by Amyotrophic Lateral Sclerosis Functional Rating Scale Revised) in the whole study population (p<0.0125), and (3) lowered neurofilament light chain (NfL) serum levels as a prognostic biomarker in the whole study population (p=0.0225).

Therefore, this study aims at prolonging survival in ALS patients by applying 1.5-fold dosage of the same intervention as in LIPCAL-ALS I in a larger number of patients, excluding patients with slow disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Possible, probable (clinically or laboratory supported) or definite amyotrophic lateral sclerosis according to the revised version of the El Escorial criteria
* Disease duration (onset of first paresis or bulbar symptoms) < 24 months
* Loss of amyotrophic lateral sclerosis functional rating scale revised of ≥ 0.33 points/month based on the formula: (48 - myotrophic lateral sclerosis functional rating scale revised score at screening visit) / (months between onset and screening visit)
* Age ≥18 years.
* Either continuously treated with a stable dose of riluzole, OR not treated with riluzole for the last 4 weeks prior to inclusion
* Either continuously treated with a stable dose of edaravone, OR not treated with edaravone for the last 4 weeks prior to inclusion
* Either continuously treated with a stable dose of sodium-phenylbutyrate/taurursodiol, OR not treated with sodium-phenylbutyrate/taurursodiol for the last 4 weeks prior to inclusion
* Capable of thoroughly understanding all information given
* full written informed consent according to good clinical practice

Exclusion Criteria:

* Previous participation in another interventional study involving an active treatment within the preceding 4 weeks
* Tracheostomy or continuous permanent ventilator dependence (>22 hours per day)
* Pregnancy or breastfeeding
* Any medical condition known to have an association with motor neuron dysfunction which might confound or obscure the diagnosis of ALS
* Presence of any concomitant life-threatening disease or impairment likely to interfere with functional assessment.
* Evidence of a major psychiatric disorder or clinically evident dementia precluding evaluation of symptoms.
* Liable to be not cooperative or comply with study requirements as assessed by the investigator, or unable to be reached in the case of emergency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Survival | 18 months
  Time from date of randomization until date of death, tracheostomy, or permanent continous ventilation (>22 hours per day)

SECONDARY OUTCOMES:
Amyotrophic Lateral Sclerosis Functional Rating Scale Revised | 18 months
  Change per month of Amyotrophic Lateral Sclerosis Functional Rating Scale Revised
Rasch Overall Amyotrophic Lateral Sclerosis Disability Scale | 18 months
  Change per month of Rasch Overall Amyotrophic Lateral Sclerosis Disability Scale
Individual Quality of Life | 18 months
  Change of Euro Quality of Life 5D 5L (EQ-5D-5L) compared to baseline
Slow vital capacity | 18 months
  Change of slow vital capacity compared to baseline
Survival | 6 months
  Time from date of randomization until date of death, tracheostomy, or permanent continous ventilation (>22 hours per day)
Survival | 12 months
  Time from date of randomization until date of death, tracheostomy, or permanent continous ventilation (>22 hours per day)
Time to death | 18 months
  Time from date of randomization until date of death
Time to tracheostomy | 18 months
  Time from date of randomization until date of tracheostomy
Time to permanent continous ventilator dependence | 18 month
  Time from date of randomization to permanent continous ventilator dependence (>22 hours per day)
Ventilation assistance-free survival | 18 months
  Time from date of randomization until implementation of mechanical ventilation
Body Mass Index | 18 months
  Change of body mass index compared to baseline
Council of Nutrition Appetite Questionnaire | 18 months
  Change of Council of Nutrition Appetite Questionnaire sum score compared to baseline
Eating Habits | 18 months
  Change of Ulm Nutrition Questionnaire compared to baseline; qualitative changes on a descriptional level (the questionnaire has no sum score); the score is meant to detect changes of eating habits and has been used in the precursor study LIPCAL-ALS I (see doi: 10.1002/ana.25661).
Neurofilament light chain | 18 months
  Change of neurofilament light chain serum levels compared to baseline
Amyotrophic Lateral Sclerosis Functional Rating Scale Revised Prediction Model | 18 months
  Difference between observed and predicted decrease of Amyotrophic Lateral Sclerosis Functional Rating Scale Revised (measured as points lost per month), based on the a prediction model, which estimates disease progression based on neurofilament light chain serum baseline levels
Neurofilament Assess Score | 18 months
  Difference between observed and predicted survival based on the Neurofilament Assess Score, a score estimating survival based on the neurofilament light chain serum baseline levels

OTHER OUTCOMES:
Microtubule-associated protein 2 in serum | 18 months
  change of Microtubule-associated protein 2 levels in serum compared to baseline
Microtubule-associated protein 2 in cerebrospinal fluid | 18 months
  change of microtubule-associated protein 2 levels in cerebrospinal fluid compared to baseline
Ubiquitin carboxy-terminal hydrolase L1 in serum | 18 months
  change of ubiquitin carboxy-terminal hydrolase L1 levels in serum compared to baseline
Ubiquitin carboxy-terminal hydrolase L1 in cerebrospinal fluid | 18 months
  change of ubiquitin carboxy-terminal hydrolase L1 levels in cerebrospinal fluid compared to baseline
Transmembrane glycoprotein NMB in serum | 18 months
  change of transmembrane glycoprotein NMB levels in serum compared to baseline
Transmembrane glycoprotein NMB in cerebrospinal fluid | 18 months
  change of transmembrane glycoprotein NMB levels in cerebrospinal fluid compared to baseline
Human cartilage glycoprotein 39 in serum | 18 months
  change of human cartilage glycoprotein 39 levels in serum compared to baseline
Human cartilage glycoprotein 39 in cerebrospinal fluid | 18 months
  change of human cartilage glycoprotein 39 levels in cerebrospinal fluid compared to baseline
SNAP-25 in serum | 18 months
  change of SNAP-25 levels in serum compared to baseline
SNAP-25 in cerebrospinal fluid | 18 months
  change of SNAP-25 levels in cerebrospinal fluid compared to baseline
Beta-synuclein in serum | 18 months
  change of beta-synuclein levels in serum compared to baseline
Beta-synuclein in cerebrospinal fluid | 18 months
  change of beta-synuclein levels in cerebrospinal fluid compared to baseline
Aquaporin-4 in serum | 18 months
  change of aquaporin-4 levels in serum compared to baseline
Aquaporin-4 in cerebrospinal fluid | 18 months
  change of aquaporin-4 levels in cerebrospinal fluid compared to baseline
Glial fibrillary acidic protein in serum | 12 months
  change of glial fibrillary acidic protein levels in serum compared to baseline
Glial fibrillary acidic protein in cerebrospinal fluid | 12 months
  change of glial fibrillary acidic protein levels in cerebrospinal fluid compared to baseline
Soluble triggering receptor expressed on myeloid cell-1 in serum | 12 months
  change of soluble triggering receptor expressed on myeloid cell-1 levels in serum compared to baseline
Soluble triggering receptor expressed on myeloid cell-1 in cerebrospinal fluid | 12 months
  change of soluble triggering receptor expressed on myeloid cell-1 levels in cerebrospinal fluid compared to baseline
CC-chemokine ligand 2 in serum | 12 months
  change of CC-chemokine ligand 2 levels in serum compared to baseline
CC-chemokine ligand 2 in cerebrospinal fluid | 12 months
  change of CC-chemokine ligand 2 levels in cerebrospinal fluid compared to baseline
interleukin-1b in serum | 12 months
  change of interleukin-1b levels in serum compared to baseline
interleukin-1b in cerebrospinal fluid | 12 months
  change of interleukin-1b levels in cerebrospinal fluid compared to baseline
interleukin-2 in serum | 12 months
  change of interleukin-2 levels in serum compared to baseline
interleukin-2 in cerebrospinal fluid | 12 months
  change of interleukin-2 levels in cerebrospinal fluid compared to baseline
interleukin-4 in serum | 12 months
  change of interleukin-4 levels in serum compared to baseline
interleukin-4 in cerebrospinal fluid | 12 months
  change of interleukin-4 levels in cerebrospinal fluid compared to baseline
interleukin-6 in serum | 12 months
  change of interleukin-6 levels in serum compared to baseline
interleukin-6 in cerebrospinal fluid | 12 months
  change of interleukin-6 levels in cerebrospinal fluid compared to baseline
interleukin-10 in serum | 12 months
  change of interleukin-10 levels in serum compared to baseline
interleukin-10 in cerebrospinal fluid | 12 months
  change of interleukin-10 levels in cerebrospinal fluid compared to baseline
interleukin-12p70 in serum | 12 months
  change of interleukin-12p70 levels in serum compared to baseline
interleukin-12p70 in cerebrospinal fluid | 12 months
  change of interleukin-12p70 levels in cerebrospinal fluid compared to baseline
interleukin-17 in serum | 12 months
  change of interleukin-17 levels in serum compared to baseline
interleukin-17 in cerebrospinal fluid | 12 months
  change of interleukin-17 levels in cerebrospinal fluid compared to baseline
Tumor necrosis factor alpha in serum | 12 months
  change of tumor necrosis factor alpha levels in serum compared to baseline
Tumor necrosis factor alpha in cerebrospinal fluid | 12 months
  change of tumor necrosis factor alpha levels in cerebrospinal fluid compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Dorst, Prof. Dr., Principal Investigator — University of Ulm
Locations (23):
- Germany (23):
  - RWTH Aachen, Aachen
  - Charité Universitätsmedizin Berlin, Berlin
  - University Clinic Bochum, Bochum
  - University Clinic Bonn, Bonn
  - Technical University Dresden, Dresden
  - University Clinic Erlangen, Erlangen
  - Alfried Krupp Krankenhaus Essen, Essen
  - University Clinic Göttingen, Göttingen
  - University Clinic Halle, Halle
  - Hannover Medical School, Hanover
  - University Clinic Jena, Jena
  - DRK Clinic Kassel, Kassel
  - Klinikum Kempten, Kempten
  - University Clinic Leipzig, Leipzig
  - University Clinic Lübeck, Lübeck
  - Diakonissenkrankenhaus Mannheim, Mannheim
  - Technical University Munich, Munich
  - University Clinic Münster, Münster
  - University Clinic Regensburg, Regensburg
  - University Clinic Rostock, Rostock
  - University of Ulm, Ulm
  - DKD HELIOS Clinic Wiesbaden, Wiesbaden
  - University Clinic Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, and figures) as well as the study protocol will be available.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 3 months and ending 5 years following article publication.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal. Data will be shared for analyses to achieve the aims in the approved proposal.
URL: https://www.uniklinik-ulm.de/neurologie.html